CLINICAL TRIAL: NCT00881075
Title: An Open-label, Baseline-Controlled Study of the Safety and Efficacy of SeeMore (TM) (EVP 1001-1 Injection) in Heart Patients
Brief Title: Safety and Efficacy of SeeMore (TM) in Heart Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eagle Vision Pharmaceutical Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1001-1:201; NCT00340925 (obsolete NCT alias)
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Myocardial Infarction
Keywords: Magnetic resonance imaging; Heart diseases; myocardial infarction; contrast agents; manganese
MeSH Terms: conditions — Myocardial Infarction; Heart Diseases | interventions — EVP 1001-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SeeMore(TM) (Experimental): intravenous imaging agent for enhanced magnetic resonance imaging.
  Interventions: Drug: SeeMore(TM)

INTERVENTIONS:
Drug: SeeMore(TM) — single dose intravenous injectable
  Other Names: EVP 1001-1

SUMMARY:
This study will examine the safety and effectiveness of a manganese-based agent called SeeMore (EVP 1001-1 Injection) for enhancing magnetic resonance imaging (MRI) in patients who have previously had a heart attack. It will determine whether SeeMore makes it easier to find damaged areas of the heart and will evaluate how well patients feel and how their bodies react after receiving the study medication.

Adult patients who have previously had a heart attack and are in stable health may be eligible for this study. Candidates are screened with a medical history, a brief physical examination and blood and urine tests.

Participants undergo the following procedures:

* Collection of blood and urine samples 24 hours before receiving SeeMore and 24 hours after. A blood sample is also taken 3 and 10 days after receiving the drug.
* MRI scans one hour before receiving SeeMore and 10 minutes after receiving the drug. MRI uses a magnetic field and radio waves to produce images of body tissues and organs. After the first (baseline) MRI is done, SeeMore is given intravenously (through a vein) and the subject's vital signs and electrocardiogram (EKG) are monitored for 10 minutes. Then the second MRI is done to determine whether the study medication makes it easier to see areas of the heart that were affected by the heart attack.
* Check of vital signs, EKG and physical examination after the second MRI.

DETAILED DESCRIPTION:
This is a Phase II open-label, baseline-controlled study. Approximately 10 adult male or nonpregnant female patients known to have had a myocardial infarct (nonacute) are intended to be enrolled at the current dose.

Prior to entry into this study, all subjects will undergo a standard physical examination including medical history, details regarding the prior myocardial infarct(s), prescription and over-the-counter drug questionnaire, vital signs, ECG, evaluation of the major organ systems, hematology, serum chemistries, and urinalysis. In addition, female subjects will undergo a serum pregnancy test. All subjects will sign an Informed Consent prior to entry into the study.

EVP 1001-1 will be administered intravenously over approximately one minute. Safety will be assessed by monitoring vital signs, ECG, and blood test after giving EVP 1001-1. MRI will be performed before and after EVP-1001-1 to measure enhancement relative to areas of myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age.
* if female, be nonpregnant as evidenced by a serum pregnancy test and using a medically-approved method of birth control, or post-menopausal or surgically sterile
* provide written informed consent after having received oral and written information about the study
* be in stable health based on medical history, examination and tests
* have potassium, calcium and hematocrit values within normal limits
* have a prior known myocardial infarction

Exclusion Criteria:

* have a positive pregnancy test (females)
* received an investigational drug or device within 30 days prior to administration of SeeMore™
* have known hypersensitivity to ondansetron or other selective serotonin 5HT3 receptor blockers
* have a history of drug abuse or alcoholism
* have had a myocardial infarct, unstable angina, stroke of transient ischemic attack (TIA) within the past six months
* are taking a digitalis preparation or calcium channel blocker
* have arrhythmias requiring medication
* have a prolonged PR interval, history of an atrioventricular conduction disorder or sick sinus syndrome
* have a prolonged QTc interval, ventricular arrhythmia or history of torsades
* have NYHA Grade III or IV heart failure
* have abnormal liver function tests or a history of liver disease
* have uncontrolled hypertension
* have potassium, calcium or hematocrit values outside normal limits
* have altered a prescription medication within 14 days or an over-the-counter medication within 7 days
* are noncompliant or otherwise unlikely to perform as required by the protocol
* if a new cardiac arrhythmia develops prior to the scheduled time for SeeMore™ administration, SeeMore™ will be withheld.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Examine the safety and tolerance of SeeMore following intravenous injection in patients known to have had a myocardial infarct | within 24 hours

SECONDARY OUTCOMES:
To assess the efficacy (enhancement features) of SeeMore for identifying myocardial infarction | within 1 hour

REFERENCES:
- [Background] Mendonca-Dias MH, Gaggelli E, Lauterbur PC. Paramagnetic contrast agents in nuclear magnetic resonance medical imaging. Semin Nucl Med. 1983 Oct;13(4):364-76. doi: 10.1016/s0001-2998(83)80048-8. PMID 6359418
- [Background] Storey P, Danias PG, Post M, Li W, Seoane PR, Harnish PP, Edelman RR, Prasad PV. Preliminary evaluation of EVP 1001-1: a new cardiac-specific magnetic resonance contrast agent with kinetics suitable for steady-state imaging of the ischemic heart. Invest Radiol. 2003 Oct;38(10):642-52. doi: 10.1097/01.rli.0000077057.88108.3f. PMID 14501492
- [Background] Storey P, Chen Q, Li W, Seoane PR, Harnish PP, Fogelson L, Harris KR, Prasad PV. Magnetic resonance imaging of myocardial infarction using a manganese-based contrast agent (EVP 1001-1): preliminary results in a dog model. J Magn Reson Imaging. 2006 Feb;23(2):228-34. doi: 10.1002/jmri.20500. PMID 16416440